CLINICAL TRIAL: NCT01820520
Title: Safety and Efficacy of Double Staining With Brilliant Blue G for Macular Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE11-09
Record Dates: First submitted 2013-03-26; First posted 2013-03-28 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Macular Hole; Epiretinal Membrane
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane | interventions — coomassie Brilliant Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Double staining with brilliant blue G during vitrectomy (Experimental)
  Interventions: Drug: brilliant blue G

INTERVENTIONS:
Drug: brilliant blue G — Double staining with brilliant blue G 0.025% for macular surgery

SUMMARY:
Study designed to evaluate the safety and efficacy of double staining with brilliant blue G 0.025% as an adjuvant to macular surgery. Patients undergoing surgery for macular hole or epiretinal membrane will be included. Safety will be evaluated by optic coherence tomography, pattern reversal electroretinogram and multifocal electroretinogram.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years of older
* Signing of informed consent
* Macular pathology requiring vitrectomy (epiretinal membrane, macular hole, vitreomacular traction syndrome)

Exclusion Criteria:

* Diagnosis of glaucoma
* Known allergy to brilliant blue G

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Thickness of ganglion cell layer - inner plexiform layer measured by optical coherence tomography | 6 months
  Average thickness of ganglion cell layer - inner plexiform layer measured by spectral domain optical coherence tomography
Amplitude of pattern reversal electroretinogram | 6 months
  Amplitude of pattern reversal electroretinogram (in microvolts)
Amplitude of b-wave of multifocal electroretinogram | 6 months
  Measurement of the amplitude of the b-wave of multifocal electroretinogram

SECONDARY OUTCOMES:
Visual acuity | 6 months
  Visual acuity measured with an Early Treatment Diabetic Retinopathy Study chart
Complications | 6 months
  Presence of any ocular complication

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico